CLINICAL TRIAL: NCT00977171
Title: An Open-Label Study To Assess The Clinical Benefit Of Droxidopa In Subjects With Chronic Fatigue Syndrome
Brief Title: Study To Assess The Clinical Benefit Of Droxidopa In Subjects With Chronic Fatigue Syndrome
Acronym: CFS201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment issues.
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Droxidopa CFS201
Record Dates: First submitted 2009-09-11; First posted 2009-09-15 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Fatigue Syndrome; Orthostatic Hypotension; Neurally Mediated Hypotension; Neurogenic Orthostatic Hypotension
Keywords: chronic fatigue syndrome; CFS; neurally mediated hypotension; NMH; neurogenic orthostatic hypotension; NOH; orthostatic hypotension; droxidopa
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Hypotension, Orthostatic | interventions — Droxidopa; 3,4-dihydroxyphenylserine aldolase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Droxidopa (Experimental)
  Interventions: Drug: Droxidopa

INTERVENTIONS:
Drug: Droxidopa — Oral, 100, 200, 300, 400, 500, or 600 mg TID, duration includes up to a 2 week titration period followed by a 12 week treatment period
  Other Names: L-threo-3,4-dihydroxyphenylserine; L-threo-DOPS; L-DOPS

SUMMARY:
A subset of patients suffering from chronic fatigue syndrome exhibit symptoms of neurally mediated hypotension. While the underlying pathophysiology of chronic fatigue syndrome is not precisely understood, a dysfunction of the autonomic nervous system is thought to play a role in this subset of patients. In several small studies, subjects within this subset have noted improvement in their chronic fatigue symptoms when treated for their neurally mediated hypotension. As droxidopa acts on the autonomic nervous system and has been shown to ameliorate symptoms of neurally mediated hypotension, it is hypothesized that droxidopa could aid in the treatment of chronic fatigue symptoms.

Neurally mediated hypotension has been associated with patients suffering from chronic fatigue syndrome. Droxidopa meanwhile has been approved in Japan for the treatment of the symptoms of neurogenic orthostatic hypotension. As such, it is hypothesized that regulating the autonomic nervous system in patients with Chronic fatigue syndrome may prove to be clinically beneficial.

DETAILED DESCRIPTION:
This is a phase II, single-center, open-label study to evaluate the efficacy and safety of droxidopa in subjects with chronic fatigue syndrome. The study will enroll enough subjects to allow 10 to be placed in the 12 week open label treatment period.

The study will consist of an initial screening period (up to 7 days) to confirm eligibility followed by an up to 2 week dose titration period, a 12 week treatment period and a 30 day follow up period to account for any new or on-going AEs. During the screening visit the following assessments will be recorded:

* Demography;
* Medical history;
* Physical examination;
* ECG;
* Vital signs (BP, HR, weight)
* Stand Test (measurement of BP and heart rate in the supine position (head and torso elevated at approximately 30° from horizontal) 10, 5, immediately before and 1, 5 and 10 minutes after standing);
* Tilt Table Test
* Blood samples for hematology and biochemistry;
* Urine sample for urinalysis
* Pregnancy test for females of child bearing potential.
* Concomitant medication review o Subjects taking ephedrine or midodrine will stop taking these drugs for at least 7 days before the baseline assessments.

Within 7 days of successful screening, the following baseline assessments will be recorded:

* Inclusion/Exclusion review;
* Standing test (measurement of BP and heart rate 10, 5, immediately before and 1, 5 and 10 minutes after standing);
* Vital signs (BP, HR, and weight);
* Urine/serum pregnancy test for WOCP;
* Concomitant medications;
* Adverse events
* Multidimensional Fatigue Inventory (MFI);
* Brief Pain Inventory (BPI);
* Clinical Global Impression of Severity (CGI-S);
* Hospital Anxiety and Depression Scale (HADS);
* Patient Global Impression of Improvement (PGI-I).

Following successful completion of screening and baseline procedures, subjects will enter the dose titration period. Subjects will be titrated upwards by 100 mg TID, preferably on consecutive days but definitely within 14 days of entry, until one of the following 3 criteria for ceasing dose escalation is met:

1. The subject has a sustained SBP of greater than 140 mmHg or DBP of greater than 90 mmHg after 1, 5 or 10 minutes of standing, OR a sustained SBP greater than 150 mmHg or DBP greater than 100 mmHg measured in the supine position (head and torso elevated at approximately 30° from horizontal).
2. The subject is unable to tolerate side effects believed to be related to the study medication;
3. The subject reaches the maximum dose of 600 mg TID droxidopa. If a subject meets criteria 1 they will proceed directly to the treatment period at the previous lower dose. Subjects meeting criteria 2 will also proceed directly to the treatment period at the previous lower dose. Subjects meeting criteria 3 will enter immediately into the treatment period at 600 mg TID.

Subjects that meet criteria 1 or 2 at the initial 100 mg TID dose will be considered baseline failures.

During treatment, the investigator can determine whether to modify the subject's dose. This determination will be based on the subject's tolerability of droxidopa.

Upon successful completion of the dose titration, subjects will begin a 12 week treatment period. Subjects will return to the clinic every 4 weeks (+/- 3 days) for efficacy, safety and compliance check. A follow-up call will occur 30 days after completion or removal of the trial to record any new or on-going AEs.

droxidopa

droxidopa [also, known as L-threo-3,4-dihydroxyphenylserine, L-threo-DOPS, or L-DOPS] is the International non-proprietary name (INN) for a synthetic amino acid precursor of norepinephrine (NE), which was originally developed by Sumitomo Pharmaceuticals Co., Limited, Japan. It has been approved for use in Japan since 1989.

Droxidopa has been shown to improve symptoms of orthostatic hypotension that result from a variety of conditions including Shy Drager syndrome (Multiple System Atrophy), Pure Autonomic Failure, and Parkinson's disease. There are four stereoisomers of DOPS; however, only the L-threo-enantiomer (droxidopa) is biologically active.

The exact mechanism of action of droxidopa in the treatment of symptomatic NOH has not been precisely defined; however, its NE replenishing properties with concomitant recovery of decreased noradrenergic activity are considered to be of major importance.

Droxidopa has been marketed in Japan since 1989. Data from clinical studies and post-marketing surveillance programs conducted in Japan show that the most commonly reported adverse drug reactions with droxidopa are increased blood pressure, nausea, and headache. In clinical studies, the prevalence and severity of droxidopa adverse effects appear to be similar to those reported by the placebo control arm.

ELIGIBILITY:
SUBJECT SELECTION CRITERIA:

* Female and male outpatients between 18-65 years of age;
* Subjects must be diagnosed with chronic fatigue syndrome (Per Fukuda Criteria);
* Subjects must have neurally mediated hypotension (NMH) or neurogenic orthostatic hypotension (NOH) (confirmed via Tilt table test);
* Voluntarily read and sign an informed consent.

MAIN SUBJECT EXCLUSION CRITERIA:

* Taking a direct acting vasoconstricting agent (i.e. ephedrine or midodrine)

  - Patients taking vasoconstrictor agents such as ephedrine, or midodrine must stop taking these drugs at least 2 days or 5 half-lives (whichever is longer) prior to their baseline visit (Visit 2);
* Taking anti-hypertensive medication for the treatment of high blood pressure
* Women of childbearing potential who are not using a medically accepted contraception;
* Subject Restrictions: Reproductive potential: Female subjects should be either post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile, or women of child-bearing potential (WOCP) who are using or agree to use acceptable methods of contraception throughout the study period and for 4 weeks after the last dose of investigational product. Acceptable contraceptives include intrauterine devices (IUDs), hormonal contraceptives (oral, depot, patch or injectable) and double barrier methods such as condoms or diaphragms with spermicidal gel or foam. If hormonal contraceptives are used they should be taken according to the package insert. WOCP who are not currently sexually active must agree to use acceptable contraception, as defined above, if they decide to become sexually active during the period of the study and for 4 weeks after the last dose of investigational product.
* For WOCP a urine pregnancy test must be conducted at screening, baseline and study termination; the results must be negative at screening and at baseline. Any positive result will be confirmed by serum beta HCG pregnancy test.
* Sexually active males whose partner is a WOCP must agree to use condoms for the duration of the study and for 4 weeks after the last dose;
* Women who are pregnant, breast feeding, or plan to become pregnant during the course of this study;
* Have a history of closed angle glaucoma;
* Have uncontrolled supine hypertension, defined as systolic blood pressure >180 mmHg and/or diastolic blood pressure >110 mmHg or use of ≥2 antihypertensive medications;
* Have atrial fibrillation or, in the investigator's opinion, have any other significant cardiac arrhythmia;
* Current melancholic major depressive disorder, or a previous diagnosis of psychosis, eating disorder, or bipolar disorder.
* History of substance abuse or dependence within the past two years, excluding nicotine and caffeine.
* Have a history of more than moderate alcohol consumption; (drinking in moderation is defined as having no more than 1 drink per day for women and no more than 2 drinks per day for men. This definition is referring to the amount consumed on any single day and is not intended as an average over several days)
* Known or suspected hypersensitivity to the study medication or any of its ingredients;
* Serious unstable medical illness, including cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other unstable medical or psychiatric conditions that in the opinion of the investigator would compromise participation or would likely lead to hospitalization during the duration of the study.
* Subjects who have acute liver injury (such as hepatitis) or severe cirrhosis (Child-Pugh Class C).
* Subjects who are judged before randomization to be at suicidal risk by the clinical investigator.
* Have diabetes mellitus or insipidus;
* Have a known or suspected current malignancy. Patients with a history of cancer must be symptom- and treatment-free for at least 5 years before randomization, with the exception of patients with non-melanoma, non-invasive skin cancers (such as basal cell carcinoma), who should not have had an intervention or recurrence within one year of starting the study;;
* Have known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug;
* In the investigator's opinion, have clinically significant abnormalities on clinical examination or laboratory testing;
* Have a serum creatinine level >1.3 mg/ml
* In the investigator's opinion, are unable to stand up without human or physical assistance;
* Conditions that Exclude a Diagnosis of CFS
* Any active medical condition that may explain the presence of chronic fatigue, such as untreated hypothyroidism, sleep apnea and narcolepsy, and iatrogenic conditions such as side effects of medication.
* Persistence of unresolved or relapsing condition that could explain the presence of chronic fatigue, Examples of illnesses that can present such a picture include some types of malignancies and chronic cases of hepatitis B or C virus infection.
* Any past or current diagnosis of a major depressive disorder with psychotic or melancholic features such as; bipolar affective disorders; schizophrenia of any subtype; delusional disorders of any subtype; dementias of any subtype; anorexia nervosa; or bulemia nervosa.
* Alcohol or other substance abuse, occurring within 2 years of the onset of chronicfatigue and any time afterwards.
* Severe obesity as defined by a body mass index [body mass index = weight in kilograms ÷ (height in meters)2] equal to or greater than 45. [Note: body mass index values vary considerably among different age groups and populations. No"normal" or "average" range of values can be suggested in a fashion that is meaningful. The BMI range of 45 or greater was selected because it clearly falls within the range of severe obesity.]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Lapp, M.D., Principal Investigator — Hunter-Hopkins Center, P.A.
Locations (1):
- 7421 Carmel Executive Park Drive, Ste. 320, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Droxidopa
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 3 patients enrolled in the study before it was stopped for difficulty recruiting subjects
Arm/Group | Droxidopa
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Impression of Improvement
Description: The CGI-I is a 7 point scale ranging from a score of 1 (very much improved) to 7 (very much worse), with no change in the middle, and assesses the improvement in relation to the baseline evaluation.
Time Frame: Baseline to end of 12 week treatment period
Population: 3 patients enrolled in the study prior to it being stopped due to difficulty enrolling patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa
Number analyzed (Participants) | 3
units on a scale | 3 (2.64)

ADVERSE EVENTS:
Arm/Group | Droxidopa
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa (N=3)
Localised infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (6)
Heart rate increased (Investigations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less